CLINICAL TRIAL: NCT05077566
Title: Immediate Exercise-Induced Hypoalgesia in Patients With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aveiro University (Other)
Responsible Party: Principal Investigator, Anabela G Silva, Assistant Professor, Aveiro University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CED8_2021
Record Dates: First submitted 2021-10-01; First posted 2021-10-14 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Oxygen Consumption

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise at 60% vo2 (Active Comparator): This arm will receive 15 minutes of exercise at 60% VO2 max.
  Interventions: Other: Exercise at 60% vo2
- Exercise at 90% vo2 (Experimental): This arm will receive 15 minutes of exercise at 90% VO2 max.
  Interventions: Other: Exercise at 90% vo2
- No intervention (No Intervention): No intervention

INTERVENTIONS:
Other: Exercise at 60% vo2 — 15 minutes of exercise at 60% VO2 max.
  Arms: Exercise at 60% vo2
Other: Exercise at 90% vo2 — 15 minutes of exercise at 90% VO2 max.
  Arms: Exercise at 90% vo2

SUMMARY:
The main objective of this study is:

• To evaluate the immediate hypoalgesic effect of an aerobic exercise session of different intensities in patients with chronic low back pain;

The secondary objective is:

• To explore whether pain intensity, level of physical activity, functionality, catastrophizing, kinesiophobia, anxiety and depression interfere with the immediate hypoalgesic effect of exercise.

DETAILED DESCRIPTION:
There will be 3 groups of participants, an asymptomatic control group that will not perform any exercise and two groups of individuals with low back pain. One group will perform exercise at 90% VO2máx and the other at 60% VO2máx.

All the three groups will be assessed at baseline for pressure pain threshold, pain intensity, pain phenotype, disability, kinesiophobia, catastrophizing, anxiety and depression, physical activity, and aerobic capacity. In addition, pressure pain threshold and pain intensity will also be assessed at post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* All groups:
* age between 18 and 65 years old
* Participants with low back pain:
* non-specific LBP (defined as pain between the costal margins and the inferior gluteal folds, which is usually accompanied by painful limitation of movement and may be associated with pain referred down to the leg)

Exclusion Criteria:

* All groups:
* presence of pathology of the nervous system, cardiovascular or carcinogenic, rheumatic diseases (for example, rheumatoid arthritis), fibromyalgia, previous history of lumbar surgery, medication that affects or alters heart rate, any contraindication to exercise and pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2021-10-03 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Pressure pain threshold | Baseline
  Pressure pain threshold measured with an algometer in Kgf
Pressure pain threshold | Post-intervention (approximately 45 minutes after baseline)
  Pressure pain threshold measured with an algometer in Kgf

SECONDARY OUTCOMES:
Aerobic capacity | Baseline
  Measured with the Chester Step Test (CST) which gives aerobic capacity and allows the calculation of percentage of VO2 max.
Physical activity | Baseline
  Measured with the International Physical Activity Questionnaire. Results can be reported in categories (low activity levels, moderate activity levels or high activity levels) or as a continuous variable (MET minutes a week).
Anxiety and depression | Baseline
  Measured with the Hospital Anxiety and Depression Scale. This scale has 2 subscales, one for Anxiety and one for Depression both scored 0 to 21 and higher values represent higher levels of anxiety and depression.
Catastrophizing | Baseline
  Measured with the Catastrophizing Scale (range 0-52 and higher values are indicative of higher pain catastrophizing)
Fear of movement | Baseline
  Measured with the TAMPA Scale of Kinesiophobia (range: 13-52 and higher values are indicative of higher levels of fear of movement)
Disability | Base
  Measured with the Roland Morris Disability Questionnaire (range: 0 to 24, with higher values indicating higher disability)
Pain phenotype | Baseline
  Measured with the Pain DETECT Scale. The final score between -1 and 38, indicates the likelihood of a neuropathic pain component. A score of ) 12 indicates that pain is unlikely to have a neuropathic component (< 15%), while a score of * 19 suggests that pain is likely to have a neuropathic component (> 90%).
Symptoms of central sensitization | Baseline
  Measured with the Central Sensitization Inventory. Score ranges from 0 to 100 and higher scores indicate higher symptoms of central sensitization.
Pain intensity | Baseline
  Assessed using the Visual Analogue Scale from 0 to 100 mm
Pain intensity | Post-intervention (approximately 45 minutes after baseline)
  Assessed using the Visual Analogue Scale from 0 to 100 mm

CONTACTS AND LOCATIONS:
Locations (1):
- Private Clinics of Physiotherapy, Aveiro, Portugal

IPD SHARING:
Plan to Share IPD: No